CLINICAL TRIAL: NCT01851148
Title: Clinical Effectiveness of Osteopathic Manipulative Treatment Versus Sham Therapy and Usual Care in Chronic Migraine: 3 Armed RCT
Brief Title: Clinical Effectiveness of Osteopathic Manipulative Treatment in Chronic Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute for Evidence Based Osteopathic Medicine (Other)
Responsible Party: Principal Investigator, Francesco Cerritelli, MS, DO, European Institute for Evidence Based Osteopathic Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MIOST-1
Record Dates: First submitted 2013-05-08; First posted 2013-05-10 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-08

CONDITIONS: Migraine
Keywords: osteopathic manipulative treatment; migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Manipulation, Osteopathic; salicylhydroxamic acid; Tryptamines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- sham therapy (Sham Comparator): subtracting serial sevel (McPartland 2003)
  Interventions: Other: sham treatment; Drug: triptans
- usual care (Other): triptans treatment only
  Interventions: Drug: triptans
- OMT (Experimental): 8 sessions of osteopathic manipulative treatment
  Interventions: Other: osteopathic manipulative treatment; Drug: triptans

INTERVENTIONS:
Other: osteopathic manipulative treatment — It consists of 8 sessions in 6 months. Each osteopathic session is based on a structural evaluation and an indirect technique treatment.
  Other Names: OMT
  Arms: OMT
Other: sham treatment — Sham therapy was administered with subjects lying supine on the treatment table while the operator used light manual contact to "treat" the subject. The practitioner's attention was distracted by subtracting serial seven calculation in silence
  Other Names: sham
  Arms: sham therapy
Drug: triptans — administration of triptans drug treatment according to international guidelines

SUMMARY:
The aim of the present study is to determine the extend to which OMT is effective on a sample of subjects affected by migraine evaluated using the headache impact test (HIT-6) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 60 years old
* chronic migraine

Exclusion Criteria:

* secondary forms of headache,
* chronic illness,
* psychiatric illness,
* post-menopausal women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2010-03; Primary Completion 2011-11 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
difference in HIT-6 score | at entry and after 26 weeks

SECONDARY OUTCOMES:
number of migraine attacks | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Cerritelli, MS, DO, Study Chair — European Institute for Evidence Based Osteopathic Medicine
Locations (1):
- Ancona's Hospital, division of neurology, Ancona, Italy

REFERENCES:
- [Result] Voigt K, Liebnitzky J, Burmeister U, Sihvonen-Riemenschneider H, Beck M, Voigt R, Bergmann A. Efficacy of osteopathic manipulative treatment of female patients with migraine: results of a randomized controlled trial. J Altern Complement Med. 2011 Mar;17(3):225-30. doi: 10.1089/acm.2009.0673. Epub 2011 Mar 8. PMID 21385086
- [Result] Schabert E, Crow WT. Impact of osteopathic manipulative treatment on cost of care for patients with migraine headache: a retrospective review of patient records. J Am Osteopath Assoc. 2009 Aug;109(8):403-7. PMID 19706829
- [Derived] Cerritelli F, Ginevri L, Messi G, Caprari E, Di Vincenzo M, Renzetti C, Cozzolino V, Barlafante G, Foschi N, Provinciali L. Clinical effectiveness of osteopathic treatment in chronic migraine: 3-Armed randomized controlled trial. Complement Ther Med. 2015 Apr;23(2):149-56. doi: 10.1016/j.ctim.2015.01.011. Epub 2015 Jan 21. PMID 25847552